CLINICAL TRIAL: NCT03722836
Title: Multicenter Observational Program Evaluation of the Efficacy and Tolerability of Detralex Treatment in Patients With Chronic Venous Edema (CEAP Class С3) in Real Clinical Practice
Brief Title: Evaluation of the Efficacy and Tolerability of Detralex in Patients With Chronic Venous Edema in Real Clinical Practice
Acronym: VAP-PRO-C3
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05682-055-RUS
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-04

CONDITIONS: Chronic Venous Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The VAP-PRO-C3 is a multicenter observational program, which is carried out in the frame of routine consultations and follow-up of patients. The program includes patients with chronic venous diseases (CVDs) of CEAP class C3. It is scheduled in Russia for 2018-2019. The program is expected to enroll 90 phlebologists from 60 cities of Russia. The planned number of patients is 900

DETAILED DESCRIPTION:
The study is aimed at evaluating the efficacy and safety of systemic pharmacotherapy (Detralex) as a part of combination treatment, and its influence on the general outcomes of treatment of patients with chronic venous edema (CEAP class C3) in real clinical practice.

Each investigator is planned to include in the program 10 patients fulfilling the inclusion criteria. The treatment will be carried out in accordance to the routine clinical practice, instructions for the medical use of drugs, and a specific clinical situation. To assess changes in edema, the method of truncated cones and duplex ultrasound scanning (DUS) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Written informed consent
* Patient did not receive treatment with venoactive drugs within the past 4 weeks prior to the inclusion in the study
* Diagnosis of chronic venous disease of class C3 (CEAP)
* Decision of an attending physician to prescribe Detralex.

Exclusion Criteria:

* Age below 18 years old
* Written informed consent is not obtained
* History of alcohol or drug abuse or use of narcotic drugs
* History of allergic reaction to diosmin or any other venoactive agent, or their intolerance
* History of allergic reaction to anesthetics and/or sclerosing agents
* Chronic venous disease of СЕАР class C0-С2 or class С4-С6
* Lymphatic edema of the lower extremities
* Secondary varicose veins, angiodysplasia, or neoplasia
* Arterial disease (ankle-brachial index <0.9)
* Infection within the past 6 weeks
* Any of the following concomitant diseases, which can affect the results:

  * Connective tissue disease (including rheumatoid arthritis), arthritis
  * Heart failure
  * Intermittent claudication (peripheral artery disease)
  * Diseases of the bones or joints of the lower extremities
  * Malignancy
* Treatment with drugs potentially causing leg edema (calcium channel blockers, hormonal drugs, NSAIDs, etc.)
* History of deep vein thrombosis (within the past year)
* History of superficial thrombophlebitis (within the past 3 months)
* Patient cannot walk (regardless of the cause)
* Obesity or body mass index [BMI] >30 kg/m2 [BMI = body mass (kg)/height (m)2]
* Predictable poor adherence to treatment
* Participation of the patient in the intervention study within the previous 3 months
* For women: pregnancy or breastfeeding, the desire to become pregnant within at least 2 months after the study
* Patient cannot attend a follow-up visit
* Patients with a contraindication to diosmin-containing agents, including Detralex

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CVD
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Stoyko, Principal Investigator
Locations (1):
- Centr of flebology, Samara, Russia

REFERENCES:
- [Derived] Bogachev VI, Boldin BV, Turkin PI, Samenkov AI; Study Group VAP-PRO-C3. [Comparative efficacy of various methods of treatment of chronic venous oedema in real clinical practice]. Angiol Sosud Khir. 2021;27(3):77-83. doi: 10.33529/ANGIO2021310. Russian. PMID 34528591

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With CVD of CEAP Class C3: the patients could receive any type of treatment for CVD
Period: Overall Study
Arm/Group | Patients With CVD of CEAP Class C3
Started | 708
Completed | 708
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With CVD of CEAP Class C3
Number analyzed (Participants) | 708
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 527
  >=65 years | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532
  Male | 176
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 708

OUTCOME MEASURES:

1. Primary Outcome: Dynamics of the Main Veno-specific Symptoms, Assessed by Visual Analog Scale (VAS) - Visit 0 vs Visit4
Description: Visual Analog Scale (VAS) was used in the VAP-PRO-C3 study in to discribe 5 criterions: 1.leg heaviness, 2.pain, 3. sensation of swelling, 4. night cramps 5. itching reduced from Description of the technique: It is a continuous scale in the form of a horizontal line 100 mm long with two extreme points located on it: "no symptom" and "the strongest symptom you can imagine." The patient is asked to place a line perpendicularly crossing the visual analogue scale at the point that corresponds to his symptom intensity. The ruler measures the distance (mm) between "no symptom" and "the strongest symptom you can imagine," providing a score range from 0 to 100. A higher score indicates a greater intensity of symptom.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients With CVD of CEAP Class C3
Number analyzed (Participants) | 708
mm
  leg heaviness- Visit 0 | 53.8 (21.9)
  leg heaviness- Visit 4 | 15.6 (15.6)
  pain- Visit 0 | 42.4 (23.9)
  pain- Visit 4 | 11.2 (13.7)
  sensation of swelling - Visit 0 | 56.8 (24.4)
  sensation of swelling - Visit 4 | 13.8 (15.9)
  night cramps -Visit 0 | 24.6 (23.3)
  night cramps -Visit 4 | 5.8 (12)
  itching -Visit 0 | 14.6 (20.6)
  itching -Visit 4 | 4.3 (10.1)

2. Primary Outcome: Changes in the Severity of Edema, as Assessed by the Method of Truncated Cones.
Description: To assess changes in edema, the method of truncated cones and duplex ultrasound scanning (DUS) will be used.
  The method is based on the assumption that the shape of the lower extremity approaches the shape of several truncated cones connected by bases that coincide in area. The volume of the cone is calculated by measuring the circumference of the upper (C) and lower (c) cones and the height (h) between them. For calculating the volume of each cone, the following formula is used:
  V = (p / 12p) ² h (C² + Cc + c²), The volume of the lower limb is determined by summing the volumes of all the cones. The smaller the height of the segments, the more accurate the result.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Patients With CVD of CEAP Class C3
Number analyzed (Participants) | 708
mL | 289 (234)

3. Secondary Outcome: Patients' Quality of Life According to CIVIQ-14 - Visit 0 vs Visit4
Description: Chronic Venous Insufficiency Questionnaire (CIVIQ-14) is a specific questionnaire for venous disease. It was used to describe the patients quality of life.
  Questionnaire consists of 3 dimenions: 1. pain in ankles or legs 2. scale of physical condition 3.influence to psychological state It is a SELF-reported survey where each patient has to circle the number (from 1 to 5): of which 1 means NO signs or symptons (the best result) and 5 stands for the worst state CIVIQ 14 consists of 14 questions, each question has a maximum score of 5 points. So 70 points indicates maximum reduced QoL, and 14 - best state of QoL.
  In order to compare the mean scores between dimensions, absolute scores were converted into an index. For each dimension, we obtained a result ranging from 0 to 100. Interpretation: the highest figure can be allocated to the lowest response option and vice versa.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: mean for index values
Arm/Group | Patients With CVD of CEAP Class C3
Number analyzed (Participants) | 708
mean for index values
  pain scale - Visit 0 | 41.0 (19.1)
  pain scale - Visit 4 | 12.8 (11.6)
  scale of physical condition -Visit 0 | 31.6 (23.8)
  scale of physical condition -Visit 4 | 11.1 (15.4)
  psychological state scale -Visit 0 | 24.5 (21.1)
  psychological state scale -Visit 4 | 5.7 (9)
  Global index score - Visit 0 | 32.4 (18.5)
  Global index score - Visit 4 | 9.9 (9.9)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Patients With CVD of CEAP Class C3
All-Cause Mortality (participants affected / at risk) | 0/708
Serious Adverse Events (participants affected / at risk) | 0/708
Other Adverse Events (participants affected / at risk) | 0/708

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03722836/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03722836/ICF_001.pdf